CLINICAL TRIAL: NCT05470036
Title: IMPRINT: A Pilot Study to Improve Germline Testing in At-Risk Patients With Prostate Cancer
Brief Title: Improving Germline Testing in At-Risk Patients With Prostate Cancer
Acronym: IMPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rana Mckay, Associate Professor of Medicine and Urology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0551
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Germline testing; Education; Video
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention (Other): In-clinic or virtual educational session on germline testing in prostate cancer with a trained educator.
  Interventions: Behavioral: Educational intervention.

INTERVENTIONS:
Behavioral: Educational intervention. — Educational intervention with trained educator on overview, rationale, implications, and risks and benefits of germline testing in prostate cancer.

SUMMARY:
A quality improvement initiative to improve rates of germline testing among men with prostate cancer through the use of an in-clinic educational session.

DETAILED DESCRIPTION:
This is a prospective single arm quality improvement initiative for the use of a standardized educational intervention on germline testing in prostate cancer to improve the rates of germline genetic testing among patients recommended for testing. Patients who consent to the study will undergo a one-on-one education session regarding the rationale and the benefits/risks of germline testing. Following the educational session, if a patient wishes to proceed with testing, they will sign the standard consent to proceed with germline testing via a commercial assay.

ELIGIBILITY:
Inclusion Criteria:

1. Men, age greater than or equal to 18 years of age.
2. Diagnosis of prostate cancer of any histology.
3. Must meet NCCN guidelines for germline testing

Exclusion Criteria:

1. Have had prior germline testing.
2. Have somatic genetic testing that is positive for a possible germline variant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rana McKay, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Video Intervention Group: All patients were enrolled to the video intervention group.
Period: Overall Study
Arm/Group | Video Intervention Group
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Education Intervention Group: In-clinic educational session on germline testing in prostate cancer with a trained educator including video intervention.
Arm/Group | Education Intervention Group
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] — Age
  years | 68 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 5
  Unknown or Not Reported | 5
Family history [Count of Participants; unit: Participants]
  No family history of cancer | 15
  Family history of cancer | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Agreeing to Proceed With Germline Testing Among Those Approached With the Educational Intervention.
Description: Germline genetic testing among adult prostate cancer patients who are recommended to receive germline testing per NCCN guidelines.
Time Frame: Within 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Educational Intervention Group: In person educational intervention group
Arm/Group | Educational Intervention Group
Number analyzed (Participants) | 50
Participants | 41

2. Secondary Outcome: Patient Baseline Knowledge of Germline Testing
Description: Assessment via baseline knowledge questionnaire.
  Survey Title: Patient Survey on Germline Testing in Prostate Cancer
  Minimum Values: 0 (No knowledge) Maximum Values: 11 (Highest knowledge)
  Higher score = higher knowledge
Time Frame: Baseline
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Education Intervention Group: All patients were enrolled to the education intervention group.
Arm/Group | Education Intervention Group
Number analyzed (Participants) | 50
Units on a scale | 9.1 [8 to 11]

3. Secondary Outcome: Patient Attitudes Towards Germline Testing and Assess the Impact of an Education Interventional on Patient Perceptions of Germline Testing
Description: Assessment via post intervention questionnaire.
  Survey Title: Patient Post-Education Patient Survey
  Minimum Values: 0 (No knowledge) Maximum Values: 11 (Highest knowledge)
  Higher score = higher knowledge
Time Frame: Within 18 months
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Education Intervention Ardm: All patients were enrolled to the education intervention group.
Arm/Group | Education Intervention Ardm
Number analyzed (Participants) | 50
Units on a scale | 9.2 [8 to 11]

4. Secondary Outcome: Number of Participants With Pathogenic Germline Mutations
Description: Assessment via tabulation of all germline pathogenic, likely pathogenic mutations and and variants of uncertain significance.
Time Frame: within 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Education Intervention Group
Number analyzed (Participants) | 50
Participants | 5

5. Secondary Outcome: Patient Knowledge of Germline Testing After the Educational Intervention.
Description: Assessment via post intervention knowledge questionnaire.
  Survey Title: Patient Survey on Germline Testing in Prostate Cancer
  Minimum Values: 0 (No knowledge) Maximum Values: 11 (Highest knowledge)
  Higher score = higher knowledge
Time Frame: within 18 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Education Intervention Group
Number analyzed (Participants) | 50
units on a scale | 9.2 [8 to 11]

ADVERSE EVENTS:
Time Frame: within 18 months
Description: Adverse events
Arm/Group | Education Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT05470036/Prot_SAP_000.pdf